CLINICAL TRIAL: NCT00957281
Title: The Association of Asthma With Systemic Inflammation and Oxidative Stress, and Its Effect on the Risk of Cardiovascular Morbidity in Adult With Stable Asthma
Brief Title: The Effect of Asthma on Systemic Inflammation, Oxidative Stress and Cardiovascular Morbidity
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Dr Ho Chung Man James, Clinical Assistant Professor, The University of Hong Kong
Other Study IDs: UW 08-306
Record Dates: First submitted 2009-08-09; First posted 2009-08-12 (Estimated); Last update posted 2009-08-12 (Estimated); Status verified 2009-08

CONDITIONS: Asthma
Keywords: Asthma; Systemic inflammation; Oxidative stress; Cardiovascular morbidity; Airway inflammation
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Plasma, serum, DNA and exhaled breath condensate
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Asthma: Asthma patients on inhaled corticosteroids

SUMMARY:
Asthma is a chronic airway inflammation which involves the interplay of different types of inflammatory cells and cytokines in the airway. The presence of systemic inflammation and oxidative stress in asthma suggests that it has a propensity to develop cardiovascular morbidity. Recent small scale studies have demonstrated that asthma severity may be associated with both airway and systemic inflammation. The investigators' study aims at linking asthma severity to airway and systemic inflammation, and subsequently to cardiovascular morbidity if a significant association of the aforementioned is present. The role of airway inflammation in contribution to systemic inflammation , and potential interaction between these two conditions will also be studied.

DETAILED DESCRIPTION:
Asthma is a chronic inflammatory airway disorder, associated with airflow obstruction and bronchial hyper-responsiveness, which affects about 10% of population in Hong Kong. It has been a major respiratory disease in Hong Kong that carries significant morbidity and high hospitalization burden in all ages. The use of long-term inhaled corticosteroid treatment in recent decades has become the cornerstone in the treatment of most patients with persistent asthma with reduction in its mortality. The ultimate goal of treatment is to achieve optimal control of airway inflammation and asthma-related mortality and morbidity.

In recent studies on the evaluation of airway and systemic inflammation in patients with asthma, various biomarkers have been measured in exhaled breath condensate (EBC), like nitric oxide, nitrates/nitrites and 8-isoprostane. Similarly, measurement of biomarkers in blood, notably high-sensitivity c-reactive protein (hs-CRP), 8-isoprostane and antioxidants (catalase, superoxide dismutase, glutathione peroxidase, glutathione), has also been used to reflect the levels of systemic inflammation and oxidative stress.

There has been substantial evidence from landmark epidemiological studies in the past 10 years, predominantly based on plasma hs-CRP, that chronic low grade systemic inflammation is an independent predictor for the development of hypertension, myocardial infarction, stroke, cardiovascular death and peripheral vascular disease. A dose-dependent risk association between hs-CRP and these cardiovascular morbidities has also been consistently demonstrated. Moreover, there has been overwhelming data to suggest the association between oxidative stress and the development cardiovascular disease. This association is easily understood in light of the cellular damages and endothelial dysfunction due to oxidative stress, which may lead to the development of atherosclerosis and cardiovascular morbidity.

In chronic obstructive pulmonary disease (COPD), a chronic inflammatory airway disorder characterized by irreversible airflow obstruction induced mainly by tobacco smoking, studies have demonstrated that, in acute exacerbations of COPD and smoking, there is a marked imbalance of redox status. The increased oxidative stress results in the inactivation of alveolar antiproteases, airspace epithelial damage, increased influx of neutrophils into lung tissue and the expression of pro-inflammatory mediators. Similarly, patients with COPD also have increase neutrophils, lymphocytes and TNF-α in the peripheral blood. In fact, many studies have demonstrated the existence of low grade systemic inflammation and oxidative stress in patients with COPD. Important studies published in recent 5 years have also linked the elevation of these systemic biomarkers, in a dose-dependent manner, to COPD severity and increased prevalence of cardiovascular and cerebrovascular morbidity and mortality in patients with COPD.

On the other hand, chronic airway inflammation is also the hallmark of asthma which involves the interplay of different types of inflammatory cells, including T-lymphocytes, eosinophils, neutrophils, macrophages and cytokines in the airway. Although the pathogenesis of asthma is incompletely understood, studies have shown that it is associated with a state of increased free radical formation, because cells derived from airways and peripheral blood of patients with asthma generate increased amount of reactive oxygen species, the level of which is related to severity of asthma. Besides, airway biomarkers indicating airway inflammation and oxidative stress have been consistently shown to be positively related to asthma severity and asthma control, which can be alleviated with treatment by inhaled corticosteroids. Additionally, recent preliminary studies have indicated that, apart from the presence of chronic airway inflammation (elevated EBC nitric oxide, EBC nitrites/nitrates and EBC 8-isoprostane), asthma may also be associated with chronic low grade systemic inflammation (elevation of plasma hs-CRP) and increased oxidative stress (increased 8-isoprostane; altered erythrocyte superoxide dismutase, catalase, glutathione peroxidase and glutathione).

Whether the presence of systemic inflammation and oxidative stress in asthma is actually a consequence of "overspill" of uncontrolled airway inflammation or the existence of an extrapulmonary source of inflammation remains unknown. At the moment, there is only little evidence on the correlation of airway and systemic inflammation in asthma, as well as the relation of systemic inflammation and oxidative stress to asthma severity. Intuitively, as in COPD, asthma-related systemic inflammation may as well increase the propensity for development of cardiovascular and cerebrovascular diseases. However, there is also a lack of study that describes the risk of cardiovascular outcomes of asthma-related systemic inflammation and oxidative stress.

Therefore, we conduct the current study with the primary objective to investigate the association of asthma severity with systemic inflammation and oxidative stress, and its effect on the risk of various cardiovascular morbidities. The secondary objective is to correlate airway inflammation and oxidative stress with systemic inflammation and oxidative stress in stable asthmatics.

ELIGIBILITY:
Inclusion Criteria:

* Asthma patients with stable persistent asthma
* Current inhaled corticosteroid users

Exclusion Criteria:

* On maintenance oral steroid
* Systemic steroid use in recent 1 month
* Asthma exacerbation (GINA criteria) in recent 1 month (ie daytime or nocturnal symptoms increment, detectable wheezing on physical examination, drop in peak flow rate, drop in spirometry indexes, increase in asthma medication, emergency medical attendance for asthma, days off work for asthma etc)
* Inhaled corticosteroid use for < 6 months
* Pregnancy

Ages: 35 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Asthma patients will be recruited from asthma clinics of 4 centres in Hong Kong, including Queen Mary Hospital, Queen Elizabeth Hospital, Kowloon Hospital and Kwong Wah Hospital.
Sampling Method: Probability Sample
Enrollment: 748 (Actual)
Dates: Start 2008-09; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Change in level of hs-CRP and oxidative stress status in relation to change in asthma severity , in terms of median, interquartile range and 95% confidence interval | 1 year

SECONDARY OUTCOMES:
Correlation coefficient of levels of EBC biomarkers with levels of hs-CRP and oxidative stress | 1 year
Interaction effect of airway inflammation on the association between asthma severity and systemic inflammation, and vice versa | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Chung-man James Ho, Principal Investigator — The University of Hong Kong
Locations (4):
- Hong Kong (4):
  - Kowloon Hospital, Hong Kong
  - Kwong Wah Hospital, Hong Kong
  - Queen Elizabeth Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong